CLINICAL TRIAL: NCT06142188
Title: A Real-world Study for the Treatment of Hematologic Malignancies With Relmacabtagene Autoleucel
Brief Title: Relmacabtagene Autoleucel in Hematologic Malignancies
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JWCAR029418
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Lymphoma, B-Cell; Large B-cell Lymphoma; Follicular Lymphoma
Keywords: Relmacabtagene Autoleucel; Chimeric antigen receptor T cells
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relmacabtagene Autoleucel: Relmacabtagene Autoleucel administered as a single IV infusion at a target dose of 1 x 10^8 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells on Day1.
  Interventions: Biological: Relmacabtagene Autoleucel

INTERVENTIONS:
Biological: Relmacabtagene Autoleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: JWCAR029

SUMMARY:
To evaluate the efficacy and safety of Relmacabtagene Autoleucel in the treatment of adult patients with hematologic malignancies in real-world

DETAILED DESCRIPTION:
The purpose of this study is to observationally evaluate the efficacy and safety data of Relmacabtagene Autoleucel for the treatment of patients with hematologic malignancies for up to 15 years after infusion. The treating physician will determine the most appropriate diagnostic and therapeutic regimen for the patient based on clinical practice. No therapeutic intervention will be administered to patients in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients who have been treated with Relma-cel, including those who have received off-label products;
3. If previously enrolled in another clinical study, they must have completed follow-up in the previous study, or have withdrawn or lost follow-up in the previous study.

Exclusion Criteria:

1.Patients who have been treated with Relma-cel and then have been treated with other CAR-T products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematologic Malignancies
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-28 (Estimated); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 15 years
  Percentage of participants with CR [CMR;CRR] or PR [partial metabolic response (PMR);

SECONDARY OUTCOMES:
CRR | 15 years
  Complete response rate
Duration of response (DOR) | 15 years
  Time from first response(PR or CR) to disease progression or death from any cause.
Progression-Free Survival (PFS) | 15 years
  PFS is defined as the time from the Relmacabtagene Autoleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Overall Survival (OS) | 15 years
  OS is defined as the time from Relmacabtagene Autoleucel infusion to the date of death from any cause.
Adverse events (AEs) | 15 years
  Types, frequency, and severity of adverse events and laboratory anomalies Physiological parameter

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No